CLINICAL TRIAL: NCT05916495
Title: An Evaluation of Remote Care (questionnaire+hybrid) in Patients Who Are Post-lung Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: patientMpower Ltd. (Industry); Manchester University NHS Foundation Trust (Other Government); University College, London (Other); New Start, The Wythenshawe Hospital Transplant Fund Centre (Unknown)
Responsible Party: Principal Investigator, John Blaikley, Senior Lecturer, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LTX patientMpower 01
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Lung Transplant; Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid care arm (Experimental): Remote review of information collected electronically will be combined with in person visits at a hospital
  Interventions: Other: Hybrid care arm
- Standard of care arm (Active Comparator): Patients will be seen in person at a hospital clinic.
  Interventions: Other: Standard of care arm

INTERVENTIONS:
Other: Hybrid care arm — Patients will be evaluated at 3 months via a remote review. This will review the patients-recorded spirometry and a questionnaire developed for this study which asses the patients' symptom burden and medication adherence. All patients participating in the study will be offered remote monitoring (patient facing app+ patient recorded home spirometry).
  Arms: Hybrid care arm
Other: Standard of care arm — Patients will be reviewed in clinic at 3 months per the standard of care. All patients participating in the study will be offered remote monitoring (patient facing app+ patient recorded home spirometry).
  Arms: Standard of care arm

SUMMARY:
Lung transplantation is used to treat patients with lung damage when there is no other treatment option. Patients require close monitoring following their transplant, with hospital check-ups every 3-4 months usually lasting all day. Although check-ups often result in no change to patient management they are essential as patients have better outcomes if complications are detected quickly.

The aim is to explore whether remote monitoring via an app (patientMpower) ± questionnaire (specifically designed to assess post-transplant patients' health), linked to a device to measure lung function, could replace some check-ups for lung transplant patients.

Patients will be randomised to receive either normal care or remote monitoring (i.e. their symptoms will be evaluated using home spirometry combined with a questionnaire). 100 lung transplant recipients will be enrolled with 50 patients being assigned to either group. Health outcomes and costs of care between the two groups will be compared

DETAILED DESCRIPTION:
100 lung transplant patients are expected to be recruited. Consent will be taken by the research team. Following admission they will be randomised to the interventional or control arms. The control arm will consist of follow-up according to unit policy, in the majority of cases this will be every 3 months. The only change is that when they come to follow up the patients will be asked to fill in the same interventional questionnaire (designed to assess post-transplant lung health) that the interventional arm are completing. However, they will be seen regardless of what this questionnaire reports.

This will act as validation for the questionnaire. The interventional arm will replace the 3 monthly visits with a questionnaire which the patient will be asked to complete and then this will be returned to the unit. The patient can fill this in via the app, or on paper and return the questionnaire via email or post. The duty clinician will then review the questionnaire and combine this with the home spirometry data which the patient is already completing to see if the patient needs to be seen. In the majority of cases, its expected that the patient will not need to be seen as the clinic visits in lung transplant are mainly monitored and the vast majority of the patients are seen every 3-4 months. Regardless of the outcome, the participant will receive a phone call from the transplant nurse within 48 hours of the appointment to discuss the results of the blood test and confirm that they are okay.

In addition to the questionnaire to assess lung health, all participants will be asked to complete other respiratory/sleep questionnaires such as Saint George's Respiratory (SGRQ), Morningness-eveningness (MEQ-SA) and the Pittsburgh Sleep Quality Index (PSQI). This will investigate whether more complex questionnaires are needed to see if patients require clinical follow-up. Study duration is predicted to be 6 months per participant. During the whole study, volunteers will be asked to wear an activity tracker such as Fitbit. Using the device's application programming interface (API) investigators will be able to remotely access data concerning heart rate, accelerometry and sleep duration, including stages of sleep. This will be accessed as required anticipated to be once per week, followed by phone calls to patients should the data be missing. In addition, their clinical record will also be accessed to obtain clinical data for instance if a sleep study has been performed. Patients will be asked to perform daily home spirometry using a Bluetooth enabled spirometer. It is currently being used in the Manchester lung transplant program. If patients have not submitted a reading for one week then they will be contacted by the study team to offer assistance.

ELIGIBILITY:
Inclusion Criteria:

* Looked after by a clinical care team at Manchester University NHS Foundation Trust
* Given consent
* Have received a lung transplant

Exclusion Criteria:

* Consent not given
* Not able to operate the remote monitoring platform

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of clinic visits per patient | 6 months
  The number of clinic follow up visits in the observation period

SECONDARY OUTCOMES:
Number of unplanned clinic visits per patient | 6 months
  The number of unplanned clinic visits in the observation period
"Measuring the Utilization Rate of Remote Monitoring for Patient Engagement" "Measuring the Utilization Rate of Remote Monitoring for Patient Engagement" Number of patient interactions with the remote monitoring platform | 6 months
  Frequency of use at ≥ 1 day/week
Hospitalisation due to deterioration of allograft function | 6 Months
  Number of patients hospitalised due to deterioration of allograft function
Duration of hospitalisations due to deterioration of allograft function | 6 Months
  Number of hospitalised days due to deterioration of allograft function
Number of planned clinic visits per patient | 6 Months
  The number of planned clinic visits in the observation period
Number of patients where symptoms were recorded accurately on the questionnaire | 6 months
  The number of patients where a clinician recorded that symptoms were recorded accuratly

CONTACTS AND LOCATIONS:
Overall Officials: John Blaikley, Principal Investigator — The University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Final results of the study will be disseminated in the form of a manuscript/s in a peer-reviewed journal scientific journals, presented at national and international conferences and in local meetings. In addition, where relevant, data from potential interim analyses will be presented at (a) relevant congress (es).

REFERENCES:
- [Derived] Varley RJ, Borton R, Van Dellen D, Santhanakrishnan K, Edwards C, Pizzo E, Blaikley JF. Description of the Protocol Investigating Whether Remote Care Can Reduce Clinic Attendance in Lung Transplantation. Pulm Ther. 2025 Dec;11(4):765-773. doi: 10.1007/s41030-025-00320-3. Epub 2025 Oct 10. PMID 41073612